CLINICAL TRIAL: NCT03542136
Title: Peripheral Neuropathy in Colorectal Cancer Patients Under Adjuvant Chemotherapy With FOLFOX, FLOX or XELOX Regime
Acronym: PENCOLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MKM-1
Record Dates: First submitted 2018-04-17; First posted 2018-05-31 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer
Keywords: Polyneuropathy; Oxaliplatin; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Polyneuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving chemotherapy treatment with oxaliplatin. (Other)
  Interventions: Device: VibrosSense Meter®

INTERVENTIONS:
Device: VibrosSense Meter® — A multi frequency tactilometry device to evaluate the vibrotactile sense to indicate the underlying (Oxaliplatin induced poly neuropathy) OIPN and then compare the results with the results of CTCAE (Common toxicity criteria of adverse events) assessment tool evaluation.

SUMMARY:
Oxaliplatin is a cytotoxic platinum compound and is one of the chemotherapeutic agent used in advanced colorectal cancer. It is used combined with Fluorouracil (5 FU) and Leucovorin. The main and most suffering side effect of oxaliplatin is polyneuropathy. Oxaliplatin-induced polyneuropathy (OIPN) can be acute and/or chronic neurotoxicity.

The early detection of the neurotoxicity and changing the medication dose and/or schedule can prevent its development. It has been used different neurotoxicity scales in grading OIPN. In this study the investigators try to investigate whether the evaluation of the vibrotactile perception VTP, by using a multi frequency tactilometry in a patients hand and foot is a good indicator and superior to the standard of care to detect the underlying OIPN in patients undergoing adjuvant chemotherapy treatment with FOLFOX, FLOX or XELOX regime.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed written informed consent.
* Fulfils the indication of the treatment with 3-6 months oxaliplatin combined adjuvant chemotherapy.
* Polyneuropathy grade according to CTCAE before treatment start ≤ 2.
* Performance status according to WHO ≤ 1.

Exclusion Criteria:

* Age < 18 years.
* The patient does not consent to the examination
* Polyneuropathy grade according to CTCAE before treatment start >2.
* Performance status according to WHO >1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of evaluating the vibrotactile sense using a multi frequency tactilometry, in patients hand and foot. This is by assessing the changes in the measurements of a multi frequency tactilometry device in between each two time points. | Investigation before cycle 1, 4, 6, 7, 8, 10, 12 and 6 months after last cycle (cycle 12), if cycle length is 2 weeks. If cycle length is 3 weeks, evaluation before cycle 1, 3, 4, 5, 6,7, 8, and 6 months after last cycle.
  Multi frequency tactilometry device is used.

SECONDARY OUTCOMES:
To evaluate if Oxaliplatin induced polyneuropathy can be earlier detected by using a multi frequency tactilometry compared with Common Terminology Criteria for Adverse Events scale (CTCAE). | Investigation before cycle 1, 4, 6, 7, 8, 10, 12 and after 6 months after last cycle (cycle 12), if cycle length is 2 weeks. If cycle length is 3 weeks, evaluation before cycle 1, 3, 4, 5, 6,7, 8, and 6 months after last cycle
  Multi frequency tactilometry device is used.

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes